CLINICAL TRIAL: NCT06528236
Title: Research on Automatic Detection of Ovarian Mass and Intelligent Auxiliary Diagnosis System Based on Multimodal Ultrasound Images
Brief Title: Research and Application of Ultrasonic Intelligent Diagnosis System for Ovarian Mass
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); Sichuan provincial maternity and child health care hospital (Unknown); The Affiliated Hospital of Qingdao University (Other); Aksu First People's Hospital (Unknown); Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024053
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Neoplasms; Adnexal Mass
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Training cohort: Training cohort is used to training artificial model based on multimodel ultrasound images or videos.
- Validation cohort: Validation cohort is used to validate artificial model.
  Interventions: Diagnostic Test: Artificial intelligence model
- Internal test cohort: Internal test cohort is used to internally test artificial model.
  Interventions: Diagnostic Test: Artificial intelligence model
- External test cohort: External test cohort is used to internally test artificial model.
  Interventions: Diagnostic Test: Artificial intelligence model

INTERVENTIONS:
Diagnostic Test: Artificial intelligence model — Using the artificial intelligence model to diagnosis benign, borderline, and malignant ovarian masses.
  Groups: External test cohort; Internal test cohort; Validation cohort

SUMMARY:
Research on automatic detection of ovarian mass and intelligent auxiliary diagnosis system based on multimodal ultrasound images.

DETAILED DESCRIPTION:
Investigators aimed to develop an ultrasonic intelligent diagnosis system for ovarian mass based on multimodal ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

1. During gynecological ultrasound examination, at least one patient with persistent ovarian tumor was found.
2. The patient underwent surgical treatment and the histopathological results.

Exclusion Criteria:

1. Histopathological analysis confirms non-ovarian tumor;
2. Histopathological results are inconclusive;
3. Issues with image quality: the ovarian mass is incomplete and does not show some surrounding tissues (but the mass is too large to exclude completely); the images are overly blurry, making it difficult to determine the characteristics of the ovarian mass (possible reasons include hardware quality issues with the ultrasound machine, motion blur, focusing problems, presence of intestinal gas in the patient); gain settings make it difficult to judge the characteristics of the ovarian mass (such as low contrast, excessively dark images, or saturation); the presence of artifacts affects the assessment of ultrasound characteristics of the ovarian mass and should be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: During gynecological ultrasound examination, at least one patient with persistent ovarian tumor was found. The patient underwent surgical treatment and the histopathological results.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve | Through study completion, an average of 1 year
  AUC (Area Under the Curve) is a common index used to evaluate the performance of binary classification model.

SECONDARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  Sensitivity refers to the ability of the test to correctly identify a positive result in an individual who actually has the disease. It represents the proportion of cases in which the test is able to detect a positive for the disease

OTHER OUTCOMES:
Specificity | Through study completion, an average of 1 year
  Specificity refers to the ability of the test to correctly identify a negative result in an individual who does not actually have the disease. It represents the proportion of cases where the disease is negative that the test is able to detect.
Accuracy | Through study completion, an average of 1 year
  Accuracy refers to the degree to which the results of the diagnostic test are consistent with the actual situation
Positive predicative value | Through study completion, an average of 1 year
  Positive Predictive Value indicates the probability that a test result will be true if it is positive. In other words, it represents the proportion of individuals who are diagnosed as positive when the test result is positive who actually have the disease
Negative predictive value | Through study completion, an average of 1 year
  Negative Predictive Value refers to the probability that if a test result is negative, the result will be true negative. It represents the proportion of individuals who are diagnosed as negative when the test results are negative that are truly free of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Litao Sun, Professor, Study Chair — Zhejiang Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No